CLINICAL TRIAL: NCT03226431
Title: Use of ARINA-1 in an Intermediate Size Patient Population of Bilateral Lung Transplant Patients With CLAD Grade 0 at Duke University to Improve FEV1
Brief Title: Use of ARINA-1 in an Intermediate Size Patient Population of Bilateral Lung Transplant Patients With CLAD Grade 0
Acronym: ARINA-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00080819
Record Dates: First submitted 2017-07-14; First posted 2017-07-21 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2018-09

CONDITIONS: Lung Transplant
MeSH Terms: interventions — Ascorbic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ARINA-1 (Experimental): Ascorbic acid (ARINA-1) (inhaled ascorbic acid 88 mg/ml) will be nebulized twice daily for 3 months using a PARI eFlow nebulizer
  Interventions: Drug: Ascorbic Acid

INTERVENTIONS:
Drug: Ascorbic Acid — ARINA-1 (inhaled ascorbic acid 88 mg/ml) will be nebulized twice daily for 3 months using a PARI eFlow nebulizer
  Other Names: ARINA-1

SUMMARY:
To treat an intermediate size patient population of bilateral lung transplant patients with CLAD-0.

DETAILED DESCRIPTION:
To treat an intermediate size patient population of bilateral lung transplant patients with CLAD-0. Treating physicians will follow standard of care for patients and monitor pulmonary function, fractional exhaled nitric oxide and quality of life of the patients.

Patient safety will be monitored by assessing changes in these parameters, as well as changes in standard of care measurements (e.g., laboratory values and x-ray images).

ELIGIBILITY:
Inclusion Criteria:

1. >6 months post-bilateral lung transplant
2. Any patient with a stable FEV1 or a decline that is < 20% from baseline.
3. No current signs of infection
4. No current signs of rejection
5. >21 years old
6. Routinely followed at the enrolling site
7. Capable of giving informed consent

Exclusion Criteria:

1. Interstitial or peribronchial/peribronchiolar fibrosis on transbronchial biopsy
2. Evidence of active congestive heart failure or symptomatic coronary artery disease, in the opinion of the site investigator
3. CLAD grade 1 or higher
4. Currently on any ICS therapy
5. Initiation of chronic azithromycin within 1 month of study enrollment (chronic azithromycin use defined as azithromycin 250mg or 500mg daily or every Monday, Wednesday, Friday)
6. Positive pregnancy test at screening, if female and of child bearing potential

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-12-11 (Actual); Primary Completion 2019-06-25 (Actual); Study Completion 2019-06-25 (Actual)

PRIMARY OUTCOMES:
Changes in FEV1 | Baseline, 1 month, 3 months, 6 months, 12 months
  Each individual's changes in pulmonary function will be assessed using the linear slope of FEV1 change from enrollment to the end of the treatment period.
Changes in FENO | Baseline
  Each individual's changes in FENO will be assessed using the change in mean baseline FENO measurements to the mean measurements post-ARINA-1 use.
Changes in Quality of Life | Baseline, 12 months
  Patient-reported quality of life measures assessed pre- and post-ARINA-1 will be compared for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Omar Mohamedaly, MD, Principal Investigator — Duke Health; Lorenzo Zaffiri, MD, Principal Investigator — Duke Health
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No